CLINICAL TRIAL: NCT00820391
Title: KIDNET vs Meditation/Relaxation - a Dissemination Randomized Controlled Treatment Trial for Children in Sri Lanka Traumatized by the War and the Tsunami
Brief Title: KIDNET Versus Meditation/Relaxation - a Dissemination RCTT for Children in Sri Lanka Traumatized by the War and the Tsunami
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: NGO vivo e.V. (Unknown); GTZ-German Technical Cooperation, rmany (Unknown); German Research Foundation (Other); Ein Herz für Kinder (Other)
Responsible Party: Dr. Claudia Catani
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: KIDNET2005
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-traumatic Stress disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KIDNET (Experimental): Narrative Exposure Therapy for Children
  Interventions: Behavioral: KIDNET
- Meditation/Relaxation (Experimental)
  Interventions: Behavioral: Meditation-Relaxation

INTERVENTIONS:
Behavioral: KIDNET — Narrative Exposure Therapy for Children - a short term intervention for the treatment of trauma after war, organized violence, torture, abuse and other detrimental life events
  Arms: KIDNET
Behavioral: Meditation-Relaxation — a protocol of traditional/local meditation and relaxation exercises, such as breathing meditation, chanting, body relaxation
  Arms: Meditation/Relaxation

SUMMARY:
The purpose of this study is to assess the efficacy of KIDNET versus a Meditation/Relaxation protocol in treating traumatized children in Sri Lanka when applied by locally trained teacher counsellors.

ELIGIBILITY:
Inclusion Criteria:

* Children with preliminary PTSD diagnosis (except for time criterion) in the age range of 8 to 14 years living in a specific IDP camp after the Tsunami disaster.

Exclusion Criteria:

* Mental retardation, psychosis, any neurological disorder

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2005-01; Primary Completion 2005-01 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Severity according to UPID; DSM IV Diagnosis of Posttraumatic Stress disorder | pre-treatment, 1 month post, 6 months follow up

SECONDARY OUTCOMES:
Functioning, Somatic Problems, School grades | pre, 1 month post, 6 months follow-up

REFERENCES:
- [Derived] Catani C, Kohiladevy M, Ruf M, Schauer E, Elbert T, Neuner F. Treating children traumatized by war and Tsunami: a comparison between exposure therapy and meditation-relaxation in North-East Sri Lanka. BMC Psychiatry. 2009 May 13;9:22. doi: 10.1186/1471-244X-9-22. PMID 19439099